CLINICAL TRIAL: NCT05086185
Title: Effect of Viscous Fiber on Postprandial Kalemic Response in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: University of Nevada, Reno (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency); Sierra Nevada Nephrology Consultants, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1596754
Record Dates: First submitted 2021-07-12; First posted 2021-10-20 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Hyperkalemia; Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: Hyperkalemia; Hemodialysis; Chronic kidney disease; Dietary fiber
MeSH Terms: conditions — Hyperkalemia; Renal Insufficiency, Chronic | interventions — Dietary Fiber

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Orange Juice (control): Orange juice providing a 0.35 mEq/kg dose of potassium
  Interventions: Diagnostic Test: Kalemic Response to Orange Juice
- Orange Juice plus Fiber: Same amount of orange juice as Orange Juice treatment with 0.15 g/kg of psyllium-based fiber added
  Interventions: Dietary Supplement: Kalemic Response to Orange Juice with Fiber

INTERVENTIONS:
Diagnostic Test: Kalemic Response to Orange Juice — 100% pulp-free orange juice
  Groups: Orange Juice (control)
Dietary Supplement: Kalemic Response to Orange Juice with Fiber — 100% pulp-free orange juice with psyllium-based fiber added
  Groups: Orange Juice plus Fiber

SUMMARY:
High blood potassium levels (hyperkalemia) is a major problem for people with kidney failure undergoing hemodialysis treatment. In order to reduce the risk of hyperkalemia, people with kidney failure are advised to limit or avoid high-potassium foods. However, high-potassium foods comprise many healthy food choices, including commonly consumed fruits and vegetables that are key sources of dietary fiber, and other important nutrients.

Risk of hyperkalemia from dietary potassium intake is most notable in the first few hours after a meal when ingested potassium enters the bloodstream. In general, dietary potassium is very well absorbed. However, dietary fiber has been shown to increase the proportion of dietary potassium that is excreted in stool. Based on these findings, it has been proposed that fiber may help to lower the risk of hyperkalemia in people with kidney disease. It remains unclear whether dietary fiber increases potassium excretion in stool by reducing the absorption of dietary potassium, or by drawing body potassium into the bowels by increasing stool bulk. The distinction may be important, as reducing potassium absorption would be expected to be of greater benefit in preventing hyperkalemia caused by eating high-potassium foods.

In this study, the investigators will assess whether a fiber supplement can reduce the effect of dietary potassium from orange juice on blood potassium levels in people with kidney disease undergoing maintenance hemodialysis treatment.

DETAILED DESCRIPTION:
The source population for this study will be adults (18-89 years old) with kidney failure undergoing thrice weekly maintenance hemodialysis (HD) treatment. Participants will include 10 patients without diabetes mellitus, and 10 patients with type 2 diabetes mellitus (T2D) that is being managed with lifestyle with or without long-acting insulin. Patients with a moderate hyperkalemia (>6.5 mEq/L) in the last 6-months, taking potassium-lowering medications, having gastrointestinal (GI) disorders that may alter potassium digestion and absorption, and low hemoglobin concentrations (<10.0 g/dL) will be excluded. In addition, participants who are deemed inappropriate for the intervention by the study Nephrologist based on cognition, prognosis or pending treatments will be excluded.

Once enrolled, participants will be asked to complete questionnaires on demographics, dietary intake, GI symptoms, and urine output. In addition, baseline data on anthropometrics, physical function, medical history and blood parameters will be obtained by physical exam and review of medical records.

Treatment measurement visits will be conducted on the same non-dialysis treatment days at the University of Nevada, Reno Clinical Research Center with participants in a fasted state. Serial blood samples will be collected before, and 60, 120 and 180 minutes after ingesting orange juice providing 0.35 mEq/kg dose of potassium alone, or with 0.15 g/kg of psyllium-based fiber. The sequence of treatments (1) orange juice or 2) orange juice + fiber) will be randomly assigned with equal allocation by T2D status. If a participant's body weight exceeds 120% of ideal body weight (IBW), then the dose of orange juice and fiber will be based on adjusted body weight.

Blood tests at times 0 and 60-minutes post-treatment will be analyzed for the basic metabolic panel plus insulin, and the 120- and 180-minutes blood samples will be analyzed for potassium concentrations. The kalemic response to study treatments will assessed based on: 1) peak change in plasma potassium concentrations, and 2) total area under the curve for plasma potassium until 180-minutes. These parameters will be compared across treatment conditions using paired t-test. If non-normally distributed, values will be log-transformed prior to analyses.

ELIGIBILITY:
Inclusion Criteria:

* Kidney failure undergoing thrice-weekly maintenance hemodialysis
* 10 patients without diabetes mellitus, and 10 patients with type 2 diabetes mellitus (T2D) that are being managed with lifestyle and/or long-acting insulin

Exclusion Criteria:

* Moderate hyperkalemia (>6.5 mEq/L) in the last 6-months.
* Potassium-lowering medications
* Gastrointestinal (GI) diseases that may alter potassium digestion and absorption.
* Low hemoglobin concentrations (<10.0 g/dL).
* Deemed to be inappropriate for the intervention by Study Nephrologist based on cognition, prognosis, or pending treatments
* Women who are pregnant or who plan to become pregnant

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population for this intervention will be adults (18-89 years) with kidney failure undergoing thrice-weekly maintenance hemodialysis treatment
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
Peak change in plasma potassium levels | 0 to 180-minutes
  The kalemic response to study treatments will be assessed based on peak change in plasma potassium concentrations compared to pre-treatment.
Plasma potassium area under the curve | 0 to 180-minutes
  The kalemic response to study treatments will be assessed based on total area under the curve for plasma potassium concentrations from pre-treatment to 180-minutes.

SECONDARY OUTCOMES:
Peak change in plasma potassium levels by diabetes status | 0 to 180-minutes
  The kalemic response to study treatments (Primary Outcome 1) will be compared between participants with and without type 2 diabetes mellitus.
Plasma potassium area under the curve by diabetes status | 0 to 180-minutes
  The kalemic response to study treatments (Primary Outcome 2) will be compared between participants with and without type 2 diabetes mellitus.

CONTACTS AND LOCATIONS:
Overall Officials: David E St-jules, PhD, Principal Investigator — University of Nevada, Reno
Locations (1):
- University of Nevada,Reno, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be available after being unidentified to those who will contact the principal investigator for research purposes.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After publishing the primary and secondary outcome paper.
Access Criteria: Anyone who is interested to do secondary analysis.

REFERENCES:
- [Background] St-Jules DE, Goldfarb DS, Sevick MA. Nutrient Non-equivalence: Does Restricting High-Potassium Plant Foods Help to Prevent Hyperkalemia in Hemodialysis Patients? J Ren Nutr. 2016 Sep;26(5):282-7. doi: 10.1053/j.jrn.2016.02.005. Epub 2016 Mar 12. PMID 26975777
- [Background] Cummings JH, Hill MJ, Jenkins DJ, Pearson JR, Wiggins HS. Changes in fecal composition and colonic function due to cereal fiber. Am J Clin Nutr. 1976 Dec;29(12):1468-73. doi: 10.1093/ajcn/29.12.1468. PMID 998555
- [Background] Allon M, Dansby L, Shanklin N. Glucose modulation of the disposal of an acute potassium load in patients with end-stage renal disease. Am J Med. 1993 May;94(5):475-482. doi: 10.1016/0002-9343(93)90081-Y. PMID 8498392